CLINICAL TRIAL: NCT06781476
Title: Evaluation of Urinary Biomarkers Trend in Preterm Very Low Birth Weight Infants: Influence of Clinical and Therapeutic Factors
Brief Title: Evaluation of Urinary Biomarkers Trend in Preterm Very Low Birth Weight Infants
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: NEO-RENE
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Kidney Injury
Keywords: kidney injury; urinary biomarkers; premature newborns

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — urinary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to define the temporal patterns of urinary biomarkers (CysC, EGF, KIM-1, NGAL, β2-Microglobulin, OPN, and MOD) in the first two weeks of life in preterm and/or very low birth weight (VLBW) infants in relation to the effect of specific factors (hsPDA, prenatal Doppler alterations) and drug therapies. Another objective is then to evaluate the predictivity of these biomarkers with respect to the occurrence of renal damage in preterm infants and possible cut-off values

DETAILED DESCRIPTION:
Premature infants represent an ever-increasing population, partly as a result of improved perinatal care in severely preterm deliveries. The prematurity condition itself and the interventions put in place in the management of this fragile category of patients can lead to even permanent changes in renal function, with potential both short-term and long-term effects (development of hypertension, chronic renal failure). The development of acute renal failure (IRA) represents one of the most frequent clinical risks, with a prevalence of 19% and an estimated incidence of 12-18%, and is an independent predictor of mortality, even after correction for potential confounding factors such as comorbidities, interventions, and demographic characteristics. This type of damage has multiple causes, including incomplete nephrogenesis, early exposure to nephrotoxic drugs, and the many nutritional problems involving the use of high-protein parenteral nutrition for long periods of time. Concomitant pathologic factors such as Botallo's duct patency, respiratory distress syndrome, and sepsis may also contribute, which may, moreover, themselves cause renal damage. It is apparent that the introduction of routine monitoring of renal function in premature infants may adiuvate the identification of infants at higher risk of developing damage and the development of individualized clinical and therapeutic approaches to safeguard the immature kidney. At present, there are no validated and established biomarkers in clinical practice for the assessment of reduced renal function in the premature infant, and often the impairment is recognized only late in life (i.e., when the ability to urinate is disrupted).

To date, the assessment of renal function in newborns has been based on the evaluation of serum creatinine: however, this analyte has proven to be a weak predictor of disease, as its levels turn out to be influenced by multiple factors such as gender, maternal renal function, age and degree of prematurity of the infant, muscle mass, current therapies, and endogenous metabolites (e.g., bilirubinemia), limiting its early predictive value with respect to the development of IRA. Creatininemia levels, moreover, do not provide specific information about the type of renal insult, and, during IRA, its changes occur later than those of estimated glomerular filtration rate (eGFR).In view of these limitations, new potential biomarkers of renal function have been investigated in order to identify molecules that can predict an early diagnosis of IRA and localize the possible site of damage, even in the subclinical phase. Among the molecules studied, the most promising currently appear to be: Cystatin C (CysC), epithelial growth factor (EGF), Neutrophil Gelatinase-Associated Lipocalin (NGAL), β2-Microglobulin, Osteopontin (OPN), kidney injury molecule 1 (KIM-1) and modulin (MOD). Important advantages of such biomarkers are the possibility of being determined noninvasively on urinary samples, without requiring additional blood samples, and the low analytical costs. In addition, the combined assessment of multiple markers could provide useful information to open new diagnostic-therapeutic perspectives in this population, shaping up as a tool to reduce short- and long-term renal morbidity. Despite promising preliminary evidence regarding the use of such markers for noninvasive serial monitoring of renal function in at-risk infants, however, further studies in the preterm population are needed before their application in normal clinical practice.

In addition, larger cohorts are needed to better assess the maturational effects of prematurity and those of other important factors, such as the presence of prenatal Doppler flowmetry alterations, on these biomarkers of renal function.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32 weeks or birth weight <1500 g;
* Admission at birth to the Neonatal Intensive Care Unit of the IRCCS A.O.U. of Bologna Policlinico di S. Orsola;
* Obtaining informed consent from parents/legal representatives.

Exclusion Criteria:

* malformations of the urinary system;
* major congenital anomalies, including congenital heart disease;
* syndromic picture or known genetic abnormalities;
* perinatal asphyxia (defined by the finding on arterial blood gas from cord blood of pH≤7.0 or base excess ≤-12 mMol/L and/or Apgar ≤5 or need for resuscitation at 10' of life);
* infants who died in the first 48 hours of life or underwent major surgery during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective cohort: number of infants enrolled in the 154/2015/U/Oss protocol. Prospective cohort: 40 patients are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Define the temporal patterns of urinary biomarkers in the first two weeks of life in preterm and/or very low birth weight infants in relation to the effect of specific factors and drug therapies | through study completion, an average of 2 year
  renal function is assessed by concentration of urinary biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Vitali, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy